CLINICAL TRIAL: NCT02174562
Title: Improving Medication Adherence in Older African Americans With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK102609-01 (NIH)
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Type 2 Diabetes; Mild Cognitive Impairment
Keywords: Type 2 diabetes; Mild Cognitive Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care-Occupational Therapy (Experimental): PC-OT consists of: 1) primary care physician (PCP) - occupational therapist (OT) collaboration; 2) DM education tailored to cognitive impairment; 3) in-home OT cognitive-functional assessment; and 4) OT-delivered Behavior Activation to increase adherence to medications and other diabetes self-management (DSM) practices (e.g., diet).
  Interventions: Behavioral: Primary Care-Occupational Therapy
- Enhanced Usual Care (Placebo Comparator): Usual care enhanced with education and controls for attention
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Primary Care-Occupational Therapy — PC-OT consists of: 1) primary care physician (PCP) - occupational therapist (OT) collaboration; 2) DM education tailored to cognitive impairment; 3) in-home OT cognitive-functional assessment; and 4) OT-delivered Behavior Activation to increase adherence to medications and other diabetes self-management (DSM) practices (e.g., diet).
  Arms: Primary Care-Occupational Therapy
Behavioral: Enhanced Usual Care — Usual care enhanced with education and attention
  Arms: Enhanced Usual Care

SUMMARY:
This research aims to help older African Americans with diabetes and mild memory problems improve how they take their medications and control their diabetes. This may preserve their independence and health, prevent cognitive and functional decline, and reduce health care costs. As the population ages and becomes more racially diverse, finding ways to achieve these outcomes has great public health importance.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes (DM) in older persons is increasing rapidly. DM increases the risk for Mild Cognitive Impairment (MCI), which is a transition state between normal cognition and dementia that is often characterized by memory and executive function deficits. These deficits reduce adherence to DM medications, which worsens glycemic control and increases the risk for adverse DM-related health outcomes. Improving medication adherence may prevent these outcomes and reduce health care costs. This is important to all older persons with DM but particularly to older African Americans (AAs). They have twice the rate of DM, worse cognitive function, lower medication adherence, and worse glycemic control than whites. One million older AAs now have DM and their number will double by 2030. Because 30% also have MCI, low medication adherence is an important problem for them. This necessitates culturally relevant interventions that compensate for their cognitive deficits and improves their medication adherence and glycemic control. We propose a randomized controlled clinical trial to test the efficacy of a collaborative Primary Care-Occupational Therapy (PC-OT) intervention to lower hemoglobin A1c (HbA1c) levels in older AAs with DM, MCI, HbA1c ≥ 7.5%, and ≤ 80% adherence to an oral hypoglycemic medication. PC-OT consists of: 1) primary care physician (PCP) - occupational therapist (OT) collaboration; 2) DM education tailored to cognitive impairment; 3) in-home OT cognitive-functional assessment; and 4) OT-delivered Behavior Activation to increase adherence to medications and other diabetes self-management (DSM) practices (e.g., diet). We will recruit 100 participants from primary care clinics and randomize them to PC-OT or Enhanced Usual Care (EUC). EUC is usual medical care plus low intensity DM education delivered by community health workers. Participants in both PC-OT and EUC will have 6 initial in-home treatment sessions over 3 months, and then 3 booster sessions during this 12 month study. The primary outcome is a reduction in HbA1c of 0.5%, which reduces the risk of adverse medical events. The primary efficacy analysis compares the proportion of participants in PC-OT and EUC who achieve this outcome at month 6 (short term effect) and at month 12 (maintenance effect). We will measure medication adherence using an electronic Medication Event Monitoring System, prescription refills, and self-reports. A secondary aim determines if improving medication adherence mediates PC-OT's impact on HbA1c levels. We will also evaluate PC-OT's effect on other DSM practices; ER visits and hospitalizations; cognition; function; mood; and quality of life; and PC-OT's costs and net financial benefits. This is the first study to determine if PCPs, collaborating with OTs (who are experts in developing strategies to compensate for cognitive/physical deficits), can improve medication adherence and glycemic control, and prevent cognitive and functional decline in older persons with DM and MCI. If PC-OT is effective in a high risk population of older AAs, its benefits may extend to all older persons with DM and have enormous public health significance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years and older.
2. Self-identified as African American, black, black American, or black/Caribbean.
3. Type II DM (i.e., physician diagnosis and medication treatment).
4. HbA1c level ≥ 7.5%.
5. MCI, based on National Institute on Aging/Alzheimer's Association (NIA/AA) criteria.
6. ≤ 80% adherence to an oral hypoglycemic medication or insuling, as documented during a run-in phase using a Medication Event Monitoring System (MEMS).

Exclusion Criteria:

1. Dementia, based on National Institute on Aging/Alzheimer's Association criteria.
2. DSM-V psychiatric disorder other than depressive disorders.
3. End-stage renal disease requiring dialysis.
4. Hearing/Vision (i.e., severe diabetic retinopathy) or motor (e.g., peripheral neuropathy) impairment that precludes research participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry W Rovner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Rovner BW, Casten RJ. Emergency department visits in African Americans with mild cognitive impairment and diabetes. J Diabetes Complications. 2021 May;35(5):107905. doi: 10.1016/j.jdiacomp.2021.107905. Epub 2021 Mar 16. PMID 33752964
- [Derived] Rovner BW, Casten RJ, Piersol CV, White N, Kelley M, Leiby BE. Improving Glycemic Control in African Americans With Diabetes and Mild Cognitive Impairment. J Am Geriatr Soc. 2020 May;68(5):1015-1022. doi: 10.1111/jgs.16339. Epub 2020 Feb 11. PMID 32043561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Care-Occupational Therapy | Enhanced Usual Care
Started | 50 | 51
Completed | 41 | 46
Not Completed | 9 | 5
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Population: A total of 101 participants with MCI were randomized to PC-OT (n = 50) or EUC (n = 51). The average age of participants was 68.4 (6.4) years (range = 60-85 years), and 62% were women. All were African American.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Care-Occupational Therapy | Enhanced Usual Care | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6.1) | 68.7 (6.7) | 68.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 19 | 19 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 50 | 51 | 101
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Improvement in Hemoglobin A1c by 0.5%"
Description: Percent of participants who had a reduction (improvement) of at least .5% in hemoglobin A1c from baseline to 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Care-Occupational Therapy | Enhanced Usual Care
Number analyzed (Participants) | 41 | 46
Participants | 25 | 22
Statistical Analysis 1: Comparison: Primary Care-Occupational Therapy vs Enhanced Usual Care; Null hypothesis is that the Relative Risk of reduction of HbA1C >=0.5 for PCOT vs EUC is 1; Test type: Superiority; p = 0.31, Poisson regression with robust SEs — 0.05 was the a priori level of significance; Risk Ratio (RR) = 1.21, 95% CI 2-sided [0.84 to 1.75] — PC-OT is the numerator, Enhanced Usual care is the denominator

2. Secondary Outcome: Adherence as Measured By Percentage of Doses Taken as Prescribed
Description: This was assessed objectively using a Medication Event Monitoring System (MEMS) bottle. The MEMS measured daily bottle openings continuously to assess adherence to insulin or an oral hypoglycemic agent. The adherence rate is the percent of doses that were taken as prescribed.
Time Frame: 4-6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of doses taken during period
Arm/Group | Primary Care-Occupational Therapy | Enhanced Usual Care
Number analyzed (Participants) | 45 | 44
percentage of doses taken during period | 61 [53 to 69] | 60 [52 to 68]
Statistical Analysis 1: Comparison: Primary Care-Occupational Therapy vs Enhanced Usual Care; Mixed effects linear regression was used to model the percentage of doses taken each month. Fixed effects were period (1-3 months, 4-6 months, 7-9 months, 10-12 months), randomization group, randomization by period interaction, stratification group, age, and run-in percentage doses taken. The outcome was transformed using the arcsin-square root transformation prior to analysis. A first-order autoregressive correlation structure was assumed; Test type: Superiority; p = 0.87, Mixed Models Analysis; P-value is for comparison of least squares means for period 2 (months 4-6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Primary Care-Occupational Therapy | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 2/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 18/50 | 16/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Care-Occupational Therapy (N=50) | Enhanced Usual Care (N=51)
Infection (Infections and infestations) | 3 (3) | 7 (12)
Cardiac events (Cardiac disorders) | 8 (9) | 4 (5)
GI (Gastrointestinal disorders) | 4 (4) | 2 (2)
Facial Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD, pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure/kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Stroke/TIA (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT02174562/Prot_SAP_001.pdf